CLINICAL TRIAL: NCT02173626
Title: Effect of Video-Module Based Mindfulness Training on Physician Stress and Well Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MultiCare Health System Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ME13.17
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Stress; Burnout; Mindfulness Skills
Keywords: Mindfulness
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSH Medical Staff (Other): Volunteers from the Good Samaritan Hospital medical staff were included on a first come first serve basis
  Interventions: Behavioral: Mindfulness Training

INTERVENTIONS:
Behavioral: Mindfulness Training — Participants enrolled on a first-come, first-serve basis, engaging in three 90-minute in person trainings, weekly online video-module trainings, and weekly teleconference coaching calls. Video-module trainings were available at all times, to be accessed at the participants' convenience. Journals and a guided meditation audio library were also provided.

SUMMARY:
An eight week mindfulness training for physicians in a community hospital setting, largely administered through web-casts, will decrease stress and burnout, increase job satisfaction, and develop lasting mindfulness skills in the participants.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the impact of a video-module based mindfulness pilot program on the stress, well-being, and mindfulness skills of physicians in a community hospital setting. We administered an eight-week mindfulness training in October/November of 2013, offered as part of a wellness initiative for medical staff in a suburban community hospital in Puyallup, Washington. Participants enrolled on a first-come, first-serve basis, engaging in three 90-minute in person trainings, weekly online video-module trainings, and weekly teleconference coaching calls. Video-module trainings were available at all times, to be accessed at the participants' convenience. Journals and a guided meditation audio library were also provided. Physician stress, well-being (emotional exhaustion, depersonalization of patients, sense of personal accomplishment), and mindfulness skills (observing, describing, acting with awareness, accepting without judgment) were evaluated at baseline, end-of-program, and eight weeks post-intervention using well-validated instruments. Risks to participants were minimal, including only the possibility of a strong emotional response to personal work undertaken by participants during the course of the study. The project was funded by MultiCare Health System.

ELIGIBILITY:
Inclusion Criteria:

* GSH medical staff member

Exclusion Criteria:

* Other MultiCare employees

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Stress | Change from baseline stress at 16 weeks
  Participant stress as measured by the Perceived Stress Scale

SECONDARY OUTCOMES:
Burnout | Change from baseline burnout at 16 weeks
  Participant well being as measured by the Maslach Burnout Inventory

OTHER OUTCOMES:
Mindfulness Skills | Change from baseline mindfulness skills at 16 weeks
  Mindfulness skills as measured by the Kentucky Inventory of Mindfulness Skills

CONTACTS AND LOCATIONS:
Overall Officials: Bethann M Pflugeisen, MS, Principal Investigator — MultiCare Health System
Locations (1):
- Good Samaritan Hospital, Puyallup, Washington, United States